CLINICAL TRIAL: NCT02606799
Title: Extracorporeal Elimination of Cytokines Following Abdominal-thoracic Esophagectomy - a Randomized Study (EXCESS)
Brief Title: Extracorporeal Elimination of Cytokines Following Abdominal-thoracic Esophagectomy
Acronym: EXCESS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No further recruitment possible due to changed conditions
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: CytoSorbents, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KIM_CS_001
Record Dates: First submitted 2015-10-01; First posted 2015-11-17 (Estimated); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Inflammation
Keywords: Esophagectomy Inflammation Hemoperfusion Cytokines
MeSH Terms: conditions — Inflammation | interventions — Hemadsorption Inhibition Tests

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (No Intervention): intensive care therapy according to international standards and following local SOPs, including fluid therapy, mechanical ventilation, catecholamine therapy and other pharmacotherapy as required
- CytoSorb (Experimental): all of the above, plus extracorporeal hemadsorption therapy (CytoSorbents Adsorber cartridge) using continuous veno-venous hemofiltration (citrate anticoagulation) CytoSorb cytokine elimination
  Interventions: Device: CytoSorb cytokine elimination

INTERVENTIONS:
Device: CytoSorb cytokine elimination — Hemoperfusion using continuous veno-venous hemofiltration (citrate regional anticoagulation) with CytoSorb cytokine elimination over a period of 48h immediately following admission to the intensive care unit
  Other Names: hemadsorption
  Arms: CytoSorb

SUMMARY:
This study evaluates the effect of extracorporeal removal of inflammatory mediators on the systemic inflammation reaction of patients admitted to the intensive care unit following elective esophagectomy. Half of the participants will be treated with an adsorption device (CytoSorbents Adsorber), while the other half will be treated according to standard care. Significant reductions of interleukin-6 plasma concentration, SOFA score and catecholamine dosage in the intervention group are expected.

DETAILED DESCRIPTION:
Radical esophagectomy combined with extensive lymphadenectomy for esophageal cancer is one of the most invasive surgical procedures. Even with progress made in surgical technique and postoperative management the rate of short- and long term complications remains high. The surgical trauma invariably causes liberation and activation of inflammatory mediators and danger associated molecular patterns, which in turn result in a pronounced systemic inflammatory reaction, leading to multiorgan dysfunction including adult respiratory distress syndrome (ARDS) in many patients. The subsequent counter regulation of the immune system induces immune paralysis, which is followed by infectious complications and increases the probability of severe sepsis. Moreover, severe systemic inflammation causes capillary leakage, resulting in impaired wound healing and endangered anastomoses.

Therefore, it seems that early and effective measures against the excessive production of mediators and cytokines are indicated without impairment of the innate and adaptive immune response as it would be expected with the administration of e.g. steroids. Instead, the removal of an excessive amount of circulating cytokines might be a desirable method having shown its effectivity in the therapy of septic shock in the past.

The aim of this study is to demonstrate the effectiveness of extracorporeal cytokine removal to dampen the systemic inflammatory response following abdominal-thoracic esophagectomy.

ELIGIBILITY:
Inclusion Criteria:

* abdominal-thoracic esophagectomy with radical lymphadenectomy
* post operative admission to ICU
* age >= 18 yrs
* written informed consent

Exclusion Criteria:

* Participation in another interventional trial
* pregnancy or lactation
* systemic medication with high dose steroids and/or immunosuppressants and/or radiotherapy during the last 3 months
* known diseases of the immune system (benign and malign)
* contraindications for extracorporeal therapy
* Thrombocytopenia < 50*10^9/l
* therapy limitations (DNR), moribund status
* missing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change of interleukin-6 plasma levels | 72 hours
  Change of interleukin-6 plasma levels

SECONDARY OUTCOMES:
Change in SOFA Score | 120 hours
  decrease of >= 2 score points in the intervention group
Change of catecholamine dose | 48 hours
  decrease of >= 0.1 µg/kg/min catecholamine dosage to achieve MAP > 65 mmHg in intervention group
Fluid intake | 120 hours
  reduction of fluid intake to maintain MAP > 65 mmHg of >= 1000 ml/24h in intervention group

CONTACTS AND LOCATIONS:
Overall Officials: Axel Nierhaus, MD, Principal Investigator — University Medical Center Hamburg-Eppendorf, Dep. of Critical Care
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Background] Panagiotou A, Gaiao S, Cruz DN. Extracorporeal therapies in sepsis. J Intensive Care Med. 2013 Sep-Oct;28(5):281-95. doi: 10.1177/0885066611425759. Epub 2011 Oct 25. PMID 22027760
- [Background] Bruenger F, Kizner L, Weile J, Morshuis M, Gummert JF. First successful combination of ECMO with cytokine removal therapy in cardiogenic septic shock: a case report. Int J Artif Organs. 2015 Feb;38(2):113-6. doi: 10.5301/ijao.5000382. Epub 2015 Feb 3. PMID 25656010
- [Background] Kellum JA, Song M, Venkataraman R. Hemoadsorption removes tumor necrosis factor, interleukin-6, and interleukin-10, reduces nuclear factor-kappaB DNA binding, and improves short-term survival in lethal endotoxemia. Crit Care Med. 2004 Mar;32(3):801-5. doi: 10.1097/01.ccm.0000114997.39857.69. PMID 15090965
- [Background] Basu R, Pathak S, Goyal J, Chaudhry R, Goel RB, Barwal A. Use of a novel hemoadsorption device for cytokine removal as adjuvant therapy in a patient with septic shock with multi-organ dysfunction: A case study. Indian J Crit Care Med. 2014 Dec;18(12):822-4. doi: 10.4103/0972-5229.146321. PMID 25538418
- [Background] Mitzner SR, Gloger M, Henschel J, Koball S. Improvement of hemodynamic and inflammatory parameters by combined hemoadsorption and hemodiafiltration in septic shock: a case report. Blood Purif. 2013;35(4):314-5. doi: 10.1159/000351206. Epub 2013 Jul 31. No abstract available. PMID 23920222
- See also: technical and scientific information — http://cytosorb-therapy.com/